CLINICAL TRIAL: NCT02363946
Title: A Double-Blind, Placebo-Controlled, Dose-Escalating, Phase 1 Study to Determine the Safety, Tolerability, Pharmacokinetics and Effect of Circulating Alpha-1 Antitrypsin Levels of ARC-AAT in Healthy Volunteer Subjects and in Patients With Alpha-1 Antitrypsin Deficiency (AATD)
Brief Title: A Study of ARC-AAT in Healthy Volunteer Subjects and Patients With Alpha-1 Antitrypsin Deficiency (AATD)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Company decision to terminate the trial
Sponsor: Arrowhead Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ARCAAT-1001; U1111-1171-0247 (Other: WHO); 2015-001147-36 (EudraCT Number)
Record Dates: First submitted 2015-02-02; First posted 2015-02-16 (Estimated); Results first posted 2018-08-03 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Alpha-1 Antitrypsin Deficiency
Keywords: alpha-1 antitrypsin; AATD
MeSH Terms: conditions — alpha 1-Antitrypsin Deficiency | interventions — Diphenhydramine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (15):
- Part A: 0.38 mg/kg (Experimental): Single dose administration of ARC-AAT intravenous (IV) injection, 0.38 mg/kg in healthy volunteers
  Interventions: Drug: ARC-AAT Injection; Drug: Diphenhydramine
- Part A: 1.0 mg/kg (Experimental): Single dose administration of ARC-AAT IV injection, 1.0 mg/kg in healthy volunteers
  Interventions: Drug: ARC-AAT Injection; Drug: Diphenhydramine
- Part A: 2.0 mg/kg (Experimental): Single dose administration of ARC-AAT IV injection, 2.0 mg/kg in healthy volunteers
  Interventions: Drug: ARC-AAT Injection; Drug: Diphenhydramine
- Part A: 3.0 mg/kg (Experimental): Single dose administration of ARC-AAT IV injection, 3.0 mg/kg in healthy volunteers
  Interventions: Drug: ARC-AAT Injection; Drug: Diphenhydramine
- Part A: 4.0 mg/kg (Experimental): Single dose administration of ARC-AAT IV injection, 4.0 mg/kg in healthy volunteers
  Interventions: Drug: ARC-AAT Injection; Drug: Diphenhydramine
- Part A: 5.0 mg/kg (Experimental): Single dose administration of ARC-AAT IV injection, 5.0 mg/kg in healthy volunteers
  Interventions: Drug: ARC-AAT Injection; Drug: Diphenhydramine
- Part A: 6.0 mg/kg (Experimental): Single dose administration of ARC-AAT IV injection, 6.0 mg/kg in healthy volunteers
  Interventions: Drug: ARC-AAT Injection; Drug: Diphenhydramine
- Part A: 7.0 mg/kg (Experimental): Single dose administration of ARC-AAT IV injection, 7.0 mg/kg in healthy volunteers
  Interventions: Drug: ARC-AAT Injection; Drug: Diphenhydramine
- Part A: 8.0 mg/kg (Experimental): Single dose administration of ARC-AAT IV injection, 8.0 mg/kg in healthy volunteers
  Interventions: Drug: ARC-AAT Injection; Drug: Diphenhydramine
- Part A: Placebo (Placebo Comparator): Single dose administration of 0.9% normal saline IV injection in healthy volunteers
  Interventions: Other: Placebo; Drug: Diphenhydramine
- Part B: 2.0 mg/kg (Experimental): Single dose administration of ARC-AAT IV injection, 2.0 mg/kg in participants with AATD
  Interventions: Drug: ARC-AAT Injection; Drug: Diphenhydramine
- Part B: 4.0 mg/kg (Experimental): Single dose administration of ARC-AAT IV injection, 4.0 mg/kg in participants with AATD
  Interventions: Drug: ARC-AAT Injection; Drug: Diphenhydramine
- Part B: 6.0 mg/kg (Experimental): Single dose administration of ARC-AAT IV injection, 6.0 mg/kg in participants with AATD
  Interventions: Drug: ARC-AAT Injection; Drug: Diphenhydramine
- Part B: 7.0 mg/kg (Experimental): Single dose administration of ARC-AAT IV injection, 7.0 mg/kg in participants with AATD
  Interventions: Drug: ARC-AAT Injection; Drug: Diphenhydramine
- Part B: Placebo (Placebo Comparator): Single dose administration of 0.9% normal saline IV injection in participants with AATD
  Interventions: Other: Placebo; Drug: Diphenhydramine

INTERVENTIONS:
Drug: ARC-AAT Injection — RNA interference-based, liver-targeted therapeutic
  Other Names: ARC-AAT
  Arms: Part A: 0.38 mg/kg; Part A: 1.0 mg/kg; Part A: 2.0 mg/kg; Part A: 3.0 mg/kg; Part A: 4.0 mg/kg; Part A: 5.0 mg/kg; Part A: 6.0 mg/kg; Part A: 7.0 mg/kg; Part A: 8.0 mg/kg; Part B: 2.0 mg/kg; Part B: 4.0 mg/kg; Part B: 6.0 mg/kg; Part B: 7.0 mg/kg
Other: Placebo — 0.9 % normal saline
  Arms: Part A: Placebo; Part B: Placebo
Drug: Diphenhydramine — Diphenhydramine 50 mg p.o. was administered 2 hours (±30 minutes) pre-dose as antihistamine pre-treatment.

SUMMARY:
The purpose of the study is to determine the safety and tolerability of escalating doses of ARC-AAT and to evaluate the pharmacokinetics of ARC-AAT and the effect of ARC-AAT on circulating levels of alpha-1 antitrypsin (AAT). The study will consist of two parts, Part A (conducted in healthy volunteers) and Part B (conducted in AATD patients) at up to 9 escalating dose levels with 6 participants per dose level.

DETAILED DESCRIPTION:
Healthy volunteers and AATD patients will be randomized to receive a single intravenous injection of either ARC-AAT or Placebo in double-blind fashion. Up to thirteen cohorts (6 participants per cohort) will be enrolled. Participants in all cohorts will be confined to the clinical facility beginning on Day -1 with discharge on Day 2. Escalation to the next dose level will proceed until a participant experiences a dose-limiting toxicity (DLT) or there is achievement of pre-determined threshold reductions in AAT levels. Dosing in participants with AATD will commence based on pre-determined threshold reductions in AAT levels for healthy volunteers. For each participant, the duration of the study clinic visits is up to 11 weeks, from Screening to the End-of-Study examination. However, including a Day 90 Follow-Up telephone call, the maximum study duration is approximately 20 weeks.

ELIGIBILITY:
Inclusion Criteria:

(Part A - Healthy Volunteers)

* Male or female healthy volunteers 18-50 years of age
* Written informed consent
* Body mass index between 18.0 and 28.0 kg/m2
* 12-lead electrocardiogram (ECG) at Screening and pre-dose assessment with no clinically significant abnormalities
* Non-pregnant/non-nursing females
* Non-smoker for at least one year with current non-smoking status confirmed by urine cotinine
* Normal lung function (or not clinically significant per investigator assessment) based on spirometry and diffusion capacity of lung for carbon monoxide (DLCO) according to American Thoracic Society (ATS) - European Respiratory Society (ERS) criteria
* Highly effective, double barrier contraception (both male and female partners) during the study and for 3 months following the dose of ARC-AAT
* Willing and able to comply with all study assessments and adhere to protocol schedule
* Suitable venous access for blood sampling
* No abnormal finding of clinical relevance at screening
* Normal AAT level

(Part B-Patients) - As for Part A with the following exceptions:

* Male or female patients 18-70 years of age
* Confirmed diagnosis of homozygous alpha 1-protease inhibitor deficiency (PiZZ genotype) not receiving alpha-1 antitrypsin augmentation therapy for more than 4 weeks
* BMI between 18.0 and 35.0 kg/m2
* Non-smoker for at least three years with current non-smoking status confirmed by urine cotinine

Exclusion Criteria:

(Part A-Healthy Volunteers)

* Current regular smoker of cigarettes or cigars or was a regular smoker over the past 1 year
* Recent (within last 6 weeks) transfusion of fresh frozen plasma, platelets, or packed red blood cells, or anticipated need for transfusion during study
* Acute signs of hepatitis/other infection within 4 weeks of screening and/or baseline
* Concurrent anticoagulants
* Use of dietary and/or herbal supplements that can interfere with liver metabolism within 7 days of screening
* Use of any drugs known to induce or inhibit hepatic drug metabolism within 14 days prior to study treatment
* Depot injection/implant of any drug other than birth control within 3 months prior to study treatment
* Diagnosis of diabetes mellitus or history of glucose intolerance
* History of poorly controlled autoimmune disease or any history of autoimmune hepatitis
* Human immunodeficiency virus (HIV) infection
* Seropositive for hepatitis B virus (HBV) or hepatitis C virus (HCV), and/or history of delta virus hepatitis
* Uncontrolled hypertension (blood pressure > 150/100 mmHg)
* History of cardiac rhythm disturbances
* Family history of congenital long QT syndrome or unexplained sudden cardiac death
* Symptomatic heart failure (per New York Heart Association [NYHA] guidelines)
* Unstable angina, myocardial infarction, severe cardiovascular disease, transient ischemic attack (TIA) or cerebrovascular accident (CVA) within past 6 months
* History of malignancy within last 5 years except adequately treated basal cell carcinoma, squamous cell skin cancer, superficial bladder tumors, or in situ cervical cancer.
* History of major surgery within 3 months of screening
* Regular use of alcohol within 1 month prior to screening (i.e., more than fourteen units of alcohol per week)
* Evidence of acute inflammation, sepsis or hemolysis or clinical evidence of lower respiratory tract infection
* Diagnosis of significant psychiatric disorder
* Use of illicit drugs (such as cocaine, phencyclidine [PCP] and crack) within 1 year prior to screening or positive urine drug screen
* History of allergy or hypersensitivity reaction to bee venom
* Use of an investigational agent or device within 30 days prior to dosing or current participation in an investigational study
* Clinically significant history/presence of any gastrointestinal pathology, unresolved gastrointestinal symptoms, liver or kidney disease
* Other conditions known to interfere with the absorption, distribution, metabolism, or excretion of drugs
* Any clinically significant history/presence of poorly controlled neurological, endocrinal, cardiovascular, pulmonary, hematological, immunologic, psychiatric, metabolic or other uncontrolled systemic disease
* Blood donation (500 mL) within 7 days prior to study treatment
* History of fever within 2 weeks of screening
* Concomitant medical/psychiatric condition or social situation that would affect compliance or result in additional safety risk
* Excessive exercise/physical activity within 3 days of screening or enrollment or planned during the study
* History of thromboembolic disease, stroke within 6 months of baseline, and/or concurrent anticoagulant medication(s)

(Part B-Patients) - As for Part A with the following exceptions:

* History of major surgery within 2 months of Screening
* Forced expiratory volume at one second (FEV1) at baseline < 60%
* AATD patients with liver elastography score > 11 at Screening

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2015-02; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- Research Site 1, Melbourne, Victoria, Australia
- Research Site 2, Homburg, Germany
- Research Site 3, Leiden, Netherlands
- Research Site 4, Edgbaston, Birmingham, United Kingdom

REFERENCES:
- [Derived] Turner AM, Stolk J, Bals R, Lickliter JD, Hamilton J, Christianson DR, Given BD, Burdon JG, Loomba R, Stoller JK, Teckman JH. Hepatic-targeted RNA interference provides robust and persistent knockdown of alpha-1 antitrypsin levels in ZZ patients. J Hepatol. 2018 Aug;69(2):378-384. doi: 10.1016/j.jhep.2018.03.012. Epub 2018 Mar 21. PMID 29572094

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study terminated early and no participants were enrolled in the 6.0 mg/kg and 7.0 mg/kg arms planned in Part B.
Groups:
- Part B: 2.0 mg/kg: Single dose administration of ARC-AAT IV injection, 2.0 mg/kg in participants with alpha-1 antitrypsin deficiency (AATD)
Period: Overall Study
Arm/Group | Part A: 0.38 mg/kg | Part A: 1.0 mg/kg | Part A: 2.0 mg/kg | Part A: 3.0 mg/kg | Part A: 4.0 mg/kg | Part A: 5.0 mg/kg | Part A: 6.0 mg/kg | Part A: 7.0 mg/kg | Part A: 8.0 mg/kg | Part A: Placebo | Part B: 2.0 mg/kg | Part B: 4.0 mg/kg | Part B: Placebo
Started | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 18 | 4 | 3 | 4
Completed | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 3 | 4 | 18 | 4 | 3 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Part A: 0.38 mg/kg: Single dose administration of ARC-AAT IV injection, 0.38 mg/kg in healthy volunteers
- Total: Total of all reporting groups
Arm/Group | Part A: 0.38 mg/kg | Part A: 1.0 mg/kg | Part A: 2.0 mg/kg | Part A: 3.0 mg/kg | Part A: 4.0 mg/kg | Part A: 5.0 mg/kg | Part A: 6.0 mg/kg | Part A: 7.0 mg/kg | Part A: 8.0 mg/kg | Part A: Placebo | Part B: 2.0 mg/kg | Part B: 4.0 mg/kg | Part B: Placebo | Total
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 18 | 4 | 3 | 4 | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.0 (9.8) | 25.0 (4.5) | 30.0 (7.8) | 29.5 (10.7) | 32.3 (5.6) | 23.8 (4.1) | 32.5 (15.3) | 26.0 (5.0) | 25.0 (1.8) | 25.4 (4.8) | 59.0 (1.8) | 64.3 (3.8) | 58.8 (9.0) | 33.4 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 2 | 1 | 1 | 4 | 3 | 3 | 2 | 12 | 3 | 1 | 3 | 40
  Male | 3 | 0 | 2 | 3 | 3 | 0 | 1 | 1 | 2 | 6 | 1 | 2 | 1 | 25

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs), or Discontinuations Due to TEAEs
Description: An adverse event (AE) is defined as any untoward medical occurrence which does not necessarily have to have a causal relationship with this treatment. TEAEs are defined as defined as AEs with onset after administration of the study drug, or when a preexisting medical condition increases in severity or frequency after study drug administration. SAEs are defined as is an AE that: results in death; is life-threatening; requires inpatient hospitalization or prolongation of an existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; is a medically important event or reaction.
Time Frame: From the first dose of study treatment through Day 29 ± 1 day
Population: All participants receiving at least 1 dose of study medication
Measure: Number; unit: participants
Arm/Group | Part A: 0.38 mg/kg | Part A: 1.0 mg/kg | Part A: 2.0 mg/kg | Part A: 3.0 mg/kg | Part A: 4.0 mg/kg | Part A: 5.0 mg/kg | Part A: 6.0 mg/kg | Part A: 7.0 mg/kg | Part A: 8.0 mg/kg | Part A: Placebo | Part B: 2.0 mg/kg | Part B: 4.0 mg/kg | Part B: Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 18 | 4 | 3 | 4
participants
  TEAEs | 2 | 2 | 2 | 1 | 3 | 3 | 3 | 1 | 3 | 9 | 3 | 2 | 4
  Study Drug Related TEAEs | 1 | 1 | 2 | 1 | 1 | 2 | 0 | 0 | 3 | 1 | 1 | 0 | 0
  Mild or Moderate TEAEs | 2 | 2 | 2 | 1 | 3 | 3 | 3 | 1 | 3 | 8 | 3 | 2 | 4
  Severe TEAEs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Study Drug Related Moderate TEAEs | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
  Study Drug Related Severe TEAEs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  SAEs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Discontinuations Due to TEAEs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Clinically Significant Treatment-Emergent Abnormalities in Laboratory Values
Description: Laboratory values collected include: hematology (haemoglobin, lymphocytes, neutrophils, platelets, white cell count, monocytes); biochemistry (alanine aminotransferase, aspartate aminotransferase, alkaline phosphatase, bilirubin, creatine kinase, creatinine, gamma-glutamyltransferase, fasting glucose, troponin I); coagulation parameters (fibrinogen, international normalized ratio); and C-reactive protein.
Time Frame: Day 1 through Day 29 ± 1 day
Population: All participants receiving at least 1 dose of study medication
Measure: Number; unit: participants
Arm/Group | Part A: 0.38 mg/kg | Part A: 1.0 mg/kg | Part A: 2.0 mg/kg | Part A: 3.0 mg/kg | Part A: 4.0 mg/kg | Part A: 5.0 mg/kg | Part A: 6.0 mg/kg | Part A: 7.0 mg/kg | Part A: 8.0 mg/kg | Part A: Placebo | Part B: 2.0 mg/kg | Part B: 4.0 mg/kg | Part B: Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 18 | 4 | 3 | 4
participants
  Troponin I | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophils | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Creatine Kinase | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White Cell Count | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Monocytes | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Red Cell Distribution Width | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

3. Primary Outcome: Number of Participants With Clinically Significant Treatment-Emergent Abnormalities in Vital Signs, Electrocardiograms (ECGs), Pulmonary Function, Physical Findings, and Other Observations
Description: Values collected include: vital signs (clinically concerning or symptomatic treatment emergent changes in heart rate, systolic blood pressure, diastolic blood pressure, respiratory rate, or temperature); ECGs (clinically significant changes from baseline were observed for ventricular rate, RR interval, QRS duration, QT interval or QT interval corrected for heart rate using Fridericia's formula [QTcF]; treatment emergent clinically significant changes in ST segments, P wave or T wave morphology; cardiac telemetry monitoring); clinically significant abnormal physical examination findings; treatment emergent sensitivity to bee venom; pulmonary function (clinically significant worsening in spirometry parameters and carbon monoxide diffusing capacity of the lung for carbon monoxide [DLCO]).
Time Frame: Day 1 through Day 29 ± 1 day
Population: All participants receiving at least 1 dose of study medication
Measure: Number; unit: participants
Arm/Group | Part A: 0.38 mg/kg | Part A: 1.0 mg/kg | Part A: 2.0 mg/kg | Part A: 3.0 mg/kg | Part A: 4.0 mg/kg | Part A: 5.0 mg/kg | Part A: 6.0 mg/kg | Part A: 7.0 mg/kg | Part A: 8.0 mg/kg | Part A: Placebo | Part B: 2.0 mg/kg | Part B: 4.0 mg/kg | Part B: Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 18 | 4 | 3 | 4
participants
  Vital Signs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  ECGs | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Physical Examination Findings | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
  Bee Venom Sensitivity | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Pulmonary Function | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

4. Primary Outcome: Pharmacokinetics of ARC-AAT: Maximum Observed Plasma Concentration (Cmax) for the Analytes AD00370 and ARC-Melittin-Like Peptide (MLP; Part A)
Time Frame: Day 1, 2, and 3 at pre-dose and then at 0.08, 0.5, 1, 3, 6, 24 and 48 hours post-dose
Population: Per protocol pharmacokinetic analysis set: all participants with evaluable concentration time profiles for each dose level who had no major protocol violations
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part A: 0.38 mg/kg | Part A: 1.0 mg/kg | Part A: 2.0 mg/kg | Part A: 3.0 mg/kg | Part A: 4.0 mg/kg | Part A: 5.0 mg/kg | Part A: 6.0 mg/kg | Part A: 7.0 mg/kg | Part A: 8.0 mg/kg
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 3
ng/mL
  Analyte AD00370 | 4430 (1175) | 15500 (2811) | 32400 (7005) | 50650 (7461) | 75625 (8152) | 93275 (6133) | 115750 (11871) | 130250 (14127) | 167000 (7810)
  Analyte ARC-MLP | 2760 (508) | 9350 (2368) | 20700 (3334) | 27050 (5390) | 43425 (3872) | 48975 (5590) | 70050 (6946) | 62525 (4029) | 84733 (2875)
Statistical Analysis 1: Comparison: Part A: 0.38 mg/kg vs Part A: 1.0 mg/kg vs Part A: 2.0 mg/kg vs Part A: 3.0 mg/kg vs Part A: 4.0 mg/kg vs Part A: 5.0 mg/kg vs Part A: 6.0 mg/kg vs Part A: 7.0 mg/kg vs Part A: 8.0 mg/kg; Dose-Proportionality of Pharmacokinetic Parameter Cmax for Analyte AD00370; Test type: Other; alpha estimate = 9.557, Standard Error of Mean 0.037 — Estimation of model: Parameter = alpha * Dose^beta. Determined from linear regression model: Log(Parameter) = log(Dose)
Statistical Analysis 2: Comparison: Part A: 0.38 mg/kg vs Part A: 1.0 mg/kg vs Part A: 2.0 mg/kg vs Part A: 3.0 mg/kg vs Part A: 4.0 mg/kg vs Part A: 5.0 mg/kg vs Part A: 6.0 mg/kg vs Part A: 7.0 mg/kg vs Part A: 8.0 mg/kg; Dose-Proportionality of Pharmacokinetic Parameter Cmax for Analyte AD00370; Test type: Other; beta estimate = 1.173, 95% CI 2-sided [1.128 to 1.218], Standard Error of Mean 0.027 — Estimation of model: Parameter = alpha * Dose^beta. Determined from linear regression model: Log(Parameter) = log(Dose); R-square (r^2)=0.98
Statistical Analysis 3: Comparison: Part A: 0.38 mg/kg vs Part A: 1.0 mg/kg vs Part A: 2.0 mg/kg vs Part A: 3.0 mg/kg vs Part A: 4.0 mg/kg vs Part A: 5.0 mg/kg vs Part A: 6.0 mg/kg vs Part A: 7.0 mg/kg vs Part A: 8.0 mg/kg; Dose-Proportionality of Pharmacokinetic Parameter Cmax for Analyte ARC-MLP; Test type: Other; alpha estimate = 9.824, Standard Error of Mean 0.030 — Estimation of model: Parameter = alpha * Dose^beta. Determined from linear regression model: Log(Parameter) = log(Dose)
Statistical Analysis 4: Comparison: Part A: 0.38 mg/kg vs Part A: 1.0 mg/kg vs Part A: 2.0 mg/kg vs Part A: 3.0 mg/kg vs Part A: 4.0 mg/kg vs Part A: 5.0 mg/kg vs Part A: 6.0 mg/kg vs Part A: 7.0 mg/kg vs Part A: 8.0 mg/kg; Dose-Proportionality of Pharmacokinetic Parameter Cmax for Analyte ARC-MLP; Test type: Other; beta estimate = 1.103, 95% CI 2-sided [1.054 to 1.153], Standard Error of Mean 0.029 — Estimation of model: Parameter = alpha * Dose^beta. Determined from linear regression model: Log(Parameter) = log(Dose); R-square (r^2)=0.98

5. Primary Outcome: Pharmacokinetics of ARC-AAT: Time to Maximum Observed Concentration (Tmax) for the Analytes AD00370 and ARC-MLP (Part A)
Time Frame: Day 1, 2, and 3 at pre-dose and then at 0.08, 0.5, 1, 3, 6, 24 and 48 hours post-dose
Population: as for outcome 4
Measure: Median (Full Range); unit: hour
Arm/Group | Part A: 0.38 mg/kg | Part A: 1.0 mg/kg | Part A: 2.0 mg/kg | Part A: 3.0 mg/kg | Part A: 4.0 mg/kg | Part A: 5.0 mg/kg | Part A: 6.0 mg/kg | Part A: 7.0 mg/kg | Part A: 8.0 mg/kg
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 3
hour
  Analyte AD00370 | 0.083 [0.083 to 0.25] | 0.083 [0.083 to 0.083] | 0.083 [0.083 to 0.083] | 0.083 [0.083 to 0.50] | 0.083 [0.083 to 0.083] | 0.083 [0.083 to 0.50] | 0.083 [0.083 to 0.50] | 0.083 [0.083 to 0.50] | 0.50 [0.083 to 0.50]
  Analyte ARC-MLP | 0.083 [0.083 to 0.25] | 0.083 [0.083 to 0.083] | 0.083 [0.083 to 0.083] | 0.083 [0.083 to 0.083] | 0.083 [0.083 to 0.50] | 0.083 [0.083 to 0.50] | 0.083 [0.083 to 1.00] | 0.50 [0.083 to 1.00] | 0.50 [0.50 to 0.50]

6. Primary Outcome: Pharmacokinetics of ARC-AAT: Area Under the Plasma Concentration Versus Time Curve From Time 0 to Time 24 Hours (AUC0-24) for the Analytes AD00370 and ARC-MLP (Part A)
Time Frame: Day 1, 2, and 3 at pre-dose and then at 0.08, 0.5, 1, 3, 6, 24 and 48 hours post-dose
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Part A: 0.38 mg/kg | Part A: 1.0 mg/kg | Part A: 2.0 mg/kg | Part A: 3.0 mg/kg | Part A: 4.0 mg/kg | Part A: 5.0 mg/kg | Part A: 6.0 mg/kg | Part A: 7.0 mg/kg | Part A: 8.0 mg/kg
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 3
hr*ng/mL
  Analyte AD00370 | 26905 (10793) | 85138 (12234) | 162198 (56129) | 282710 (61810) | 438532 (38111) | 541628 (49787) | 708648 (212442) | 763392 (96095) | 908117 (144892)
  Analyte ARC-MLP | 28734 (6757) | 82627 (32332) | 213250 (67886) | 291876 (58240) | 458790 (48790) | 459939 (81820) | 699833 (85172) | 716938 (46783) | 1011569 (101693)
Statistical Analysis 1: Comparison: Part A: 0.38 mg/kg vs Part A: 1.0 mg/kg vs Part A: 2.0 mg/kg vs Part A: 3.0 mg/kg vs Part A: 4.0 mg/kg vs Part A: 5.0 mg/kg vs Part A: 6.0 mg/kg vs Part A: 7.0 mg/kg vs Part A: 8.0 mg/kg; Dose-Proportionality of Pharmacokinetic Parameter AUC0-24 for Analyte AD00370; Test type: Other; alpha estimate = 11.274, Standard Error of Mean 0.057 — Estimation of model: Parameter = alpha * Dose^beta. Determined from linear regression model: Log(Parameter) = log(Dose)
Statistical Analysis 2: Comparison: Part A: 0.38 mg/kg vs Part A: 1.0 mg/kg vs Part A: 2.0 mg/kg vs Part A: 3.0 mg/kg vs Part A: 4.0 mg/kg vs Part A: 5.0 mg/kg vs Part A: 6.0 mg/kg vs Part A: 7.0 mg/kg vs Part A: 8.0 mg/kg; Dose-Proportionality of Pharmacokinetic Parameter AUC0-24 for Analyte AD00370; Test type: Other; beta estimate = 1.181, 95% CI 2-sided [1.112 to 1.249], Standard Error of Mean 0.040 — Estimation of model: Parameter = alpha * Dose^beta. Determined from linear regression model: Log(Parameter) = log(Dose); R-square (r^2)=0.96
Statistical Analysis 3: Comparison: Part A: 0.38 mg/kg vs Part A: 1.0 mg/kg vs Part A: 2.0 mg/kg vs Part A: 3.0 mg/kg vs Part A: 4.0 mg/kg vs Part A: 5.0 mg/kg vs Part A: 6.0 mg/kg vs Part A: 7.0 mg/kg vs Part A: 8.0 mg/kg; Dose-Proportionality of Pharmacokinetic Parameter AUC0-24 for Analyte ARC-MLP; Test type: Other; alpha estimate = 12.133, Standard Error of Mean 0.040 — Estimation of model: Parameter = alpha * Dose^beta. Determined from linear regression model: Log(Parameter) = log(Dose)
Statistical Analysis 4: Comparison: Part A: 0.38 mg/kg vs Part A: 1.0 mg/kg vs Part A: 2.0 mg/kg vs Part A: 3.0 mg/kg vs Part A: 4.0 mg/kg vs Part A: 5.0 mg/kg vs Part A: 6.0 mg/kg vs Part A: 7.0 mg/kg vs Part A: 8.0 mg/kg; Dose-Proportionality of Pharmacokinetic Parameter AUC0-24 for Analyte ARC-MLP; Test type: Other; beta estimate = 1.147, 95% CI 2-sided [1.080 to 1.215], Standard Error of Mean 0.040 — Estimation of model: Parameter = alpha * Dose^beta. Determined from linear regression model: Log(Parameter) = log(Dose); R-square (r^2)=0.96

7. Primary Outcome: Pharmacokinetics of ARC-AAT: Area Under the Plasma Concentration Versus Time Curve From From Zero to Infinity (AUCinf) for the Analytes AD00370 and ARC-MLP (Part A)
Time Frame: Day 1, 2, and 3 at pre-dose and then at 0.08, 0.5, 1, 3, 6, 24 and 48 hours post-dose
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Part A: 0.38 mg/kg | Part A: 1.0 mg/kg | Part A: 2.0 mg/kg | Part A: 3.0 mg/kg | Part A: 4.0 mg/kg | Part A: 5.0 mg/kg | Part A: 6.0 mg/kg | Part A: 7.0 mg/kg | Part A: 8.0 mg/kg
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 3
hr*ng/mL
  Analyte AD00370 | 27388 (11183) | 85906 (12529) | 164856 (58070) | 285487 (62310) | 441239 (39032) | 547045 (52126) | 719843 (226599) | 771924 (100469) | 916343 (147924)
  Analyte ARC-MLP | 34718 (8345) | 103116 (48837) | 277684 (119873) | 380506 (89117) | 559372 (82769) | 569056 (129569) | 872798 (136277) | 952668 (99324) | 1251318 (138571)
Statistical Analysis 1: Comparison: Part A: 0.38 mg/kg vs Part A: 1.0 mg/kg vs Part A: 2.0 mg/kg vs Part A: 3.0 mg/kg vs Part A: 4.0 mg/kg vs Part A: 5.0 mg/kg vs Part A: 6.0 mg/kg vs Part A: 7.0 mg/kg vs Part A: 8.0 mg/kg; Dose-Proportionality of Pharmacokinetic Parameter AUCinf for Analyte AD00370; Test type: Other; alpha estimate = 11.286, Standard Error of Mean 0.058 — Estimation of model: Parameter = alpha * Dose^beta. Determined from linear regression model: Log(Parameter) = log(Dose)
Statistical Analysis 2: Comparison: Part A: 0.38 mg/kg vs Part A: 1.0 mg/kg vs Part A: 2.0 mg/kg vs Part A: 3.0 mg/kg vs Part A: 4.0 mg/kg vs Part A: 5.0 mg/kg vs Part A: 6.0 mg/kg vs Part A: 7.0 mg/kg vs Part A: 8.0 mg/kg; Dose-Proportionality of Pharmacokinetic Parameter AUCinf for Analyte AD00370; Test type: Other; beta estimate = 1.179, 95% CI 2-sided [1.110 to 1.249], Standard Error of Mean 0.041 — Estimation of model: Parameter = alpha * Dose^beta. Determined from linear regression model: Log(Parameter) = log(Dose); R-square (r^2)=0.96
Statistical Analysis 3: Comparison: Part A: 0.38 mg/kg vs Part A: 1.0 mg/kg vs Part A: 2.0 mg/kg vs Part A: 3.0 mg/kg vs Part A: 4.0 mg/kg vs Part A: 5.0 mg/kg vs Part A: 6.0 mg/kg vs Part A: 7.0 mg/kg vs Part A: 8.0 mg/kg; Dose-Proportionality of Pharmacokinetic Parameter AUCinf for Analyte ARC-MLP; Test type: Other; alpha estimate = 12.347, Standard Error of Mean 0.049 — Estimation of model: Parameter = alpha * Dose^beta. Determined from linear regression model: Log(Parameter) = log(Dose)
Statistical Analysis 4: Comparison: Part A: 0.38 mg/kg vs Part A: 1.0 mg/kg vs Part A: 2.0 mg/kg vs Part A: 3.0 mg/kg vs Part A: 4.0 mg/kg vs Part A: 5.0 mg/kg vs Part A: 6.0 mg/kg vs Part A: 7.0 mg/kg vs Part A: 8.0 mg/kg; Dose-Proportionality of Pharmacokinetic Parameter AUCinf for Analyte ARC-MLP; Test type: Other; beta estimate = 1.163, 95% CI 2-sided [1.081 to 1.245], Standard Error of Mean 0.049 — Estimation of model: Parameter = alpha * Dose^beta. Determined from linear regression model: Log(Parameter) = log(Dose); R-square (r^2)=0.95

8. Primary Outcome: Pharmacokinetics of ARC-AAT: Terminal Elimination Rate Constant Obtained From the Slope of the Line (Kel) for the Analytes AD00370 and ARC-MLP (Part A)
Time Frame: Day 1, 2, and 3 at pre-dose and then at 0.08, 0.5, 1, 3, 6, 24 and 48 hours post-dose
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: 1/hour
Arm/Group | Part A: 0.38 mg/kg | Part A: 1.0 mg/kg | Part A: 2.0 mg/kg | Part A: 3.0 mg/kg | Part A: 4.0 mg/kg | Part A: 5.0 mg/kg | Part A: 6.0 mg/kg | Part A: 7.0 mg/kg | Part A: 8.0 mg/kg
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 3
1/hour
  Analyte AD00370 | 0.186 (0.050) | 0.177 (0.004) | 0.170 (0.013) | 0.174 (0.004) | 0.185 (0.011) | 0.183 (0.006) | 0.185 (0.023) | 0.178 (0.010) | 0.181 (0.009)
  Analyte ARC-MLP | 0.0786 (0.0141) | 0.0879 (0.0297) | 0.0778 (0.0265) | 0.0762 (0.0218) | 0.0846 (0.0158) | 0.0815 (0.0231) | 0.0768 (0.0104) | 0.0622 (0.0077) | 0.0730 (0.0046)

9. Primary Outcome: Pharmacokinetics of ARC-AAT: Half-Life (t1/2) for the Analytes AD00370 and ARC-MLP (Part A)
Time Frame: Day 1, 2, and 3 at pre-dose and then at 0.08, 0.5, 1, 3, 6, 24 and 48 hours post-dose
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Part A: 0.38 mg/kg | Part A: 1.0 mg/kg | Part A: 2.0 mg/kg | Part A: 3.0 mg/kg | Part A: 4.0 mg/kg | Part A: 5.0 mg/kg | Part A: 6.0 mg/kg | Part A: 7.0 mg/kg | Part A: 8.0 mg/kg
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 3
hours
  Analyte AD00370 | 3.90 (0.84) | 3.91 (0.09) | 4.09 (0.31) | 3.99 (0.09) | 3.75 (0.22) | 3.78 (0.12) | 3.80 (0.53) | 3.90 (0.23) | 3.83 (0.19)
  Analyte ARC-MLP | 9.02 (1.50) | 8.60 (2.88) | 9.77 (3.39) | 9.83 (3.46) | 8.43 (1.68) | 8.93 (1.98) | 9.17 (1.40) | 11.3 (1.5) | 9.52 (0.61)

10. Primary Outcome: Percentage Reduction From Baseline of AAT Up to Day 29
Description: Clinical assay for total serum AAT level was used for Part A. A quantitative measurement of AAT was used for Part B. A negative percent reduction indicates a percentage increase. Baseline AAT levels consisted of a geometric mean based on 3 assessments taken prior to study drug administration: at 2 time points during the Screening window at least 5 days apart, and on Day -1.
Time Frame: Baseline, Days 3, 8, 15, 22 and 29
Population: All participants who received a full dose of study drug with evaluable data at given time point.
Measure: Mean (Standard Deviation); unit: percentage reduction
Arm/Group | Part A: 0.38 mg/kg | Part A: 1.0 mg/kg | Part A: 2.0 mg/kg | Part A: 3.0 mg/kg | Part A: 4.0 mg/kg | Part A: 5.0 mg/kg | Part A: 6.0 mg/kg | Part A: 7.0 mg/kg | Part A: 8.0 mg/kg | Part A: Placebo | Part B: 2.0 mg/kg | Part B: 4.0 mg/kg | Part B: Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 3 | 18 | 3 | 3 | 4
percentage reduction
  Day 3: number analyzed (Participants) | 4 | 4 | 4 | 3 | 4 | 4 | 4 | 4 | 3 | 18 | 3 | 3 | 4
  Day 3 | -4.70 (8.45) | -7.00 (3.19) | -1.94 (4.49) | 13.76 (4.74) | 20.76 (5.86) | 21.65 (5.28) | 22.20 (8.80) | 20.35 (11.83) | 30.07 (6.37) | -4.65 (11.13) | 11.5 (11.5) | 43.8 (5.6) | -13.0 (31.9)
  Day 8: number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 3 | 3 | 18 | 3 | 3 | 4
  Day 8 | 0.93 (2.86) | 10.90 (8.30) | 13.40 (11.68) | 33.20 (14.33) | 46.92 (6.16) | 58.52 (6.15) | 58.44 (7.50) | 50.95 (6.82) | 58.66 (2.99) | -0.26 (10.80) | 43.1 (26.7) | 54.4 (22.2) | 7.0 (36.9)
  Day 15: number analyzed (Participants) | 4 | 4 | 4 | 3 | 4 | 4 | 4 | 3 | 3 | 17 | 3 | 3 | 4
  Day 15 | 5.00 (2.62) | 3.89 (2.78) | 26.72 (14.31) | 33.65 (14.66) | 61.53 (11.75) | 74.20 (7.03) | 75.75 (5.95) | 73.57 (2.76) | 79.18 (4.03) | 0.78 (11.91) | 37.5 (20.4) | 77.7 (1.5) | 7.2 (19.8)
  Day 22: number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 3 | 3 | 17 | 3 | 3 | 4
  Day 22 | 1.42 (4.01) | 6.81 (8.81) | 15.59 (9.21) | 35.50 (15.24) | 58.64 (13.55) | 77.18 (9.94) | 83.12 (3.67) | 81.14 (1.17) | 87.47 (2.09) | 0.50 (13.48) | 25.1 (17.2) | 59.5 (13.4) | 1.7 (20.8)
  Day 29: number analyzed (Participants) | 4 | 4 | 4 | 3 | 4 | 4 | 4 | 4 | 3 | 18 | 3 | 3 | 4
  Day 29 | 0.19 (10.37) | 25.87 (6.58) | 13.93 (17.16) | 27.40 (10.65) | 50.02 (20.46) | 73.15 (14.46) | 82.99 (4.19) | 78.20 (7.83) | 87.93 (1.75) | -1.56 (8.66) | 21.0 (24.4) | 65.2 (8.7) | -7.2 (30.3)

11. Secondary Outcome: Number of Participants With AAT Reduction > 30% From Baseline (First Occurrence)
Description: Data presents the study visit day upon which a participant had the first occurrence of AAT reduction of > 30% from Baseline, and the number of participants who had a > 30% reduction at any visit (overall). Baseline AAT levels consisted of a geometric mean based on 3 assessments taken prior to study drug administration: at 2 time points during the Screening window at least 5 days apart, and on Day -1.
Time Frame: Baseline, Days 3, 8, 15, 22 and 29
Population: All participants who received a full dose of study drug with evaluable data at given time point.
Measure: Number; unit: participants
Arm/Group | Part A: 0.38 mg/kg | Part A: 1.0 mg/kg | Part A: 2.0 mg/kg | Part A: 3.0 mg/kg | Part A: 4.0 mg/kg | Part A: 5.0 mg/kg | Part A: 6.0 mg/kg | Part A: 7.0 mg/kg | Part A: 8.0 mg/kg | Part A: Placebo | Part B: 2.0 mg/kg | Part B: 4.0 mg/kg | Part B: Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 3 | 18 | 3 | 3 | 4
participants
  Overall | 0 | 2 | 2 | 3 | 4 | 4 | 4 | 4 | 3 | 0 | 2 | 3 | 1
  Day 3 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 3 | 0
  Day 8 | 0 | 0 | 0 | 1 | 4 | 4 | 3 | 2 | 1 | 0 | 2 | 0 | 1
  Day 15 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 22 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Day 29 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

12. Secondary Outcome: Maximum Percentage Reduction in Mean AAT (Nadir of Mean AAT)
Time Frame: Study Day for Nadir of Mean AAT: Day 8 (for Part B 2 mg/kg arm), Day 15 (for Part A 0.38 mg/kg, 2 mg/kg, 4 mg/ kg, Placebo arms; Part B 4 mg/kg, Placebo arms), Day 22 (Part A 3 mg/kg, 5 mg/kg, 6 mg/kg, 7 mg/kg arms), Day 29 (1 mg/kg, 8 mg/kg arms)
Population: All participants who received a full dose of study drug.
Measure: Number; unit: percentage reduction
Arm/Group | Part A: 0.38 mg/kg | Part A: 1.0 mg/kg | Part A: 2.0 mg/kg | Part A: 3.0 mg/kg | Part A: 4.0 mg/kg | Part A: 5.0 mg/kg | Part A: 6.0 mg/kg | Part A: 7.0 mg/kg | Part A: 8.0 mg/kg | Part A: Placebo | Part B: 2.0 mg/kg | Part B: 4.0 mg/kg | Part B: Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 3 | 18 | 3 | 3 | 4
percentage reduction | 5.0 | 25.9 | 26.7 | 35.5 | 61.5 | 77.2 | 83.1 | 81.1 | 87.9 | 0.78 | 43.1 | 77.7 | 7.2

13. Secondary Outcome: Number of Participants With a Return From Nadir AAT Blood Levels to Above Normal or Within 15% of Baseline in > 100 Days
Description: Baseline AAT levels consisted of a geometric mean based on 3 assessments taken prior to study drug administration: at 2 time points during the Screening window at least 5 days apart, and on Day -1.
Time Frame: Baseline, up to Day 29, and through 100 days of follow-up
Population: All participants
Measure: Number; unit: participants
Arm/Group | Part A: 0.38 mg/kg | Part A: 1.0 mg/kg | Part A: 2.0 mg/kg | Part A: 3.0 mg/kg | Part A: 4.0 mg/kg | Part A: 5.0 mg/kg | Part A: 6.0 mg/kg | Part A: 7.0 mg/kg | Part A: 8.0 mg/kg | Part A: Placebo | Part B: 2.0 mg/kg | Part B: 4.0 mg/kg | Part B: Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 18 | 4 | 3 | 4
participants | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 18 | 4 | 3 | 4

14. Secondary Outcome: Mean Percentage Change in Circulating Blood Levels of Cytokines 2 Hours Post-Dose
Time Frame: Pre-dose, 2 hours post-dose
Population: Participants with available data for given parameter.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Part A: 0.38 mg/kg | Part A: 1.0 mg/kg | Part A: 2.0 mg/kg | Part A: 3.0 mg/kg | Part A: 4.0 mg/kg | Part A: 5.0 mg/kg | Part A: 6.0 mg/kg | Part A: 7.0 mg/kg | Part A: 8.0 mg/kg | Part A: Placebo | Part B: 2.0 mg/kg | Part B: 4.0 mg/kg | Part B: Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 18 | 4 | 1 | 3
percentage change
  Serum interleukin-1 beta | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | -9 (17) | 9 (18) | 0 (0) | -2 (10) | 114 (NA) — only 1 participant evaluated | 0 (0)
  Serum interleukin-6 | 5 (8) | 79 (141) | 95 (113) | 50 (64) | 277 (308) | 100 (191) | 146 (261) | 258 (285) | 364 (255) | -1 (7) | 60 (52) | 130 (NA) — only 1 participant evaluated | 56 (91)
  Serum interleukin-8 | 32 (70) | 280 (328) | 336 (297) | 103 (101) | 1712 (981) | 564 (576) | 252 (363) | 695 (635) | 2015 (1569) | -6 (17) | 197 (319) | 46 (NA) — only 1 participant evaluated | -44 (13)
  Serum interleukin-10 | -5 (19) | 72 (134) | 51 (52) | 42 (45) | 27 (54) | 19 (28) | 116 (160) | 377 (498) | 638 (536) | -2 (7) | 0 (0) | 0 (NA) — only 1 participant evaluated | -5 (8)
  Serum interleukin-12p40 | 2 (37) | 2 (5) | 5 (8) | 6 (9) | 0 (0) | 0 (0) | 152 (217) | -9 (19) | 29 (38) | -3 (10) | -4 (13) | 79 (NA) — only 1 participant evaluated | 0 (0)
  Serum interleukin-12p70 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 54 (108) | 0 (0) | 0 (0) | 166 (389) | 82 (130) | -1 (4) | -3 (5) | 48 (NA) — only 1 participant evaluated | 23 (40)
  Serum monocyte chemoattractant protein-1 | 123 (171) | 442 (133) | 505 (254) | 632 (281) | 1176 (427) | 1297 (747) | 543 (497) | 906 (720) | 2014 (427) | 1 (13) | 262 (262) | 44 (NA) — only 1 participant evaluated | -27 (14)
  Serum macrophage inflammatory protein-1 alpha | 147 (126) | 294 (275) | 386 (556) | 264 (438) | 1674 (1022) | 1096 (578) | 406 (416) | 1003 (814) | 854 (538) | 15 (69) | 246 (304) | 0 (NA) — only 1 participant evaluated | 0 (0)
  Serum tumor necrosis factor alpha | 66 (69) | 207 (90) | 286 (90) | 187 (156) | 818 (344) | 476 (137) | 301 (237) | 761 (492) | 742 (273) | 3 (27) | 107 (152) | 55 (NA) — only 1 participant evaluated | -29 (11)
  Serum interferon alpha 2 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (7) | 73 (147) | 172 (366) | 515 (529) | 5 (20) | -3 (7) | 700 (NA) — only 1 participant evaluated | 69 (119)

15. Secondary Outcome: Mean Percentage Change in Circulating Blood Levels of Complement Factors 2 Hours Post-Dose
Time Frame: Pre-dose, 2 hours post-dose
Population: Participants with available data for given parameter.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Part A: 0.38 mg/kg | Part A: 1.0 mg/kg | Part A: 2.0 mg/kg | Part A: 3.0 mg/kg | Part A: 4.0 mg/kg | Part A: 5.0 mg/kg | Part A: 6.0 mg/kg | Part A: 7.0 mg/kg | Part A: 8.0 mg/kg | Part A: Placebo | Part B: 2.0 mg/kg | Part B: 4.0 mg/kg | Part B: Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 4 | 18 | 4 | 1 | 3
percentage change
  Plasma Bb | 18 (16) | 56 (25) | 76 (37) | 133 (29) | 181 (185) | 137 (85) | 70 (63) | 147 (73) | 309 (174) | -7 (9) | 56 (61) | 59 (NA) — only 1 participant evaluated | -14 (7)
  Serum C3a | -12 (6) | 30 (42) | -22 (24) | -0 (8) | 71 (156) | -5 (18) | 14 (56) | 40 (50) | 34 (30) | -11 (23) | -18 (23) | 219 (NA) — only 1 participant evaluated | 16 (40)
  Serum C4a | -5 (7) | 37 (70) | -11 (10) | 2 (8) | 16 (13) | -8 (27) | 78 (107) | 60 (53) | -1 (15) | -19 (35) | -35 (21) | 160 (NA) — only 1 participant evaluated | -15 (42)
  Serum C5a | 2 (7) | 2 (7) | -16 (5) | -2 (25) | -14 (7) | 2 (15) | 0 (8) | 6 (6) | 6 (12) | -2 (18) | -4 (16) | 22 (NA) — only 1 participant evaluated | -4 (10)
  Serum CH50 | -5 (8) | -14 (11) | -14 (7) | -8 (8) | -16 (4) | -17 (8) | -10 (4) | -13 (13) | -19 (10) | -3 (9) | -3 (3) | -18 (NA) — only 1 participant evaluated | -0 (13)

ADVERSE EVENTS:
Time Frame: Day -1 through Day 29 ± 1 day
Arm/Group | Part A: 0.38 mg/kg | Part A: 1.0 mg/kg | Part A: 2.0 mg/kg | Part A: 3.0 mg/kg | Part A: 4.0 mg/kg | Part A: 5.0 mg/kg | Part A: 6.0 mg/kg | Part A: 7.0 mg/kg | Part A: 8.0 mg/kg | Part A: Placebo | Part B: 2.0 mg/kg | Part B: 4.0 mg/kg | Part B: Placebo
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4 | 0/4 | 0/4 | 0/4 | 0/4 | 0/4 | 0/4 | 0/4 | 0/18 | 0/4 | 0/3 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/4 | 0/4 | 0/4 | 0/4 | 0/4 | 0/4 | 0/4 | 1/18 | 0/4 | 0/3 | 0/4
Other Adverse Events (participants affected / at risk) | 2/4 | 2/4 | 2/4 | 1/4 | 3/4 | 3/4 | 3/4 | 1/4 | 3/4 | 9/18 | 3/4 | 2/3 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: 0.38 mg/kg (N=4) | Part A: 1.0 mg/kg (N=4) | Part A: 2.0 mg/kg (N=4) | Part A: 3.0 mg/kg (N=4) | Part A: 4.0 mg/kg (N=4) | Part A: 5.0 mg/kg (N=4) | Part A: 6.0 mg/kg (N=4) | Part A: 7.0 mg/kg (N=4) | Part A: 8.0 mg/kg (N=4) | Part A: Placebo (N=18) | Part B: 2.0 mg/kg (N=4) | Part B: 4.0 mg/kg (N=3) | Part B: Placebo (N=4)
Rhabdomyolosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A: 0.38 mg/kg (N=4) | Part A: 1.0 mg/kg (N=4) | Part A: 2.0 mg/kg (N=4) | Part A: 3.0 mg/kg (N=4) | Part A: 4.0 mg/kg (N=4) | Part A: 5.0 mg/kg (N=4) | Part A: 6.0 mg/kg (N=4) | Part A: 7.0 mg/kg (N=4) | Part A: 8.0 mg/kg (N=4) | Part A: Placebo (N=18) | Part B: 2.0 mg/kg (N=4) | Part B: 4.0 mg/kg (N=3) | Part B: Placebo (N=4)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tension headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral coldness (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeling cold (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Troponin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No